CLINICAL TRIAL: NCT06326970
Title: SPECT Fibroblast Activation Protein Imaging in Patients With Cardiac Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Other Study IDs: HenanICE202401
Record Dates: First submitted 2024-03-09; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 99mTc-FAPI imaging in heart diseases: Participant involves patients with myocarditis, hypertension, arrhythmia, myocardial infarction, dilated cardiomyopathy, and cardiac tumors.
  Interventions: Diagnostic Test: 99mTc-FAPI SPECT imaging

INTERVENTIONS:
Diagnostic Test: 99mTc-FAPI SPECT imaging — 99mTc radionuclide is labeled to a HYINC-FAPI-04 probe as a tracer. SPECT imaging was performed 2 hours after 99mTc-FAPI intravenous injection into the subject, and image processing and quantitative analysis were performed using the Q.Volumetrix MI System software package.

SUMMARY:
This observational study aims to learn about the preliminary exploration of 99mTc-FAPI imaging in heart diseases and its potential application.

Participant involves patients with myocarditis, pulmonary hypertension, arrhythmia, myocardial infarction, dilated cardiomyopathy, and cardiac tumors, health conditions may also studied as control.

The main questions it aims to answer are 1, radionuclide 99mTc labeled fibroblast-activated protein inhibitors (99mTc-FAPI) imaging in the use of cardiac diseases and its limitations. 2, the performance in subjects with different control of hypertension to evaluate myocardial injury and fibrosis for providing a molecular biological basis for the study of diseases and mechanisms.

Participants will undergo 99mTc-FAPI imaging by Single-photon emission computed tomography (SPECT) and record their cardiac disease characterization and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis or suspected of cardiac injury
* Must be able to receive PET/CT scan

Exclusion Criteria:

* Pregnant women
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or confirmed myocarditis, pulmonary hypertension, arrhythmia, myocardial infarction, dilated cardiomyopathy, and cardiac tumors.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
positive uptake | 3 months
  99mTc-FAPI accumulation on the heart, measure the standardized uptake values (SUV)

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, Ph.D., Principal Investigator — Fuwai central China hospital; Jing Cui, Ph.D., Principal Investigator — Fuwai central China hospital

IPD SHARING:
Plan to Share IPD: No